CLINICAL TRIAL: NCT01695772
Title: A Multi-Center, Single-Arm, Pilot Study of 5-FU Based Doublet Chemotherapy Plus Bevacizumab as Neoadjuvant Therapy for Patients With Previously Untreated Unresectable Liver-Only Metastases From Colorectal Cancer
Brief Title: A Study of Bevacizumab Plus 5-Flurouracil (5-FU) Based Doublet Chemotherapy as Neoadjuvant Therapy for Participants With Previously Untreated Unresectable Liver-Only Metastases From Colorectal Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28419
Record Dates: First submitted 2012-09-27; First posted 2012-09-28 (Estimated); Results first posted 2016-07-28 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Bevacizumab (Experimental)
  Interventions: Drug: 5-FU based doublet chemotherapy; Drug: bevacizumab

INTERVENTIONS:
Drug: 5-FU based doublet chemotherapy — Standard 5-FU based doublet chemotherapy. Protocol did not specify any particular chemotherapy regimen. The choice of 5-FU based doublet chemotherapy was as per standard of practice and the dosage of 5-FU based doublet chemotherapy was as per product labels.
Drug: bevacizumab — 5 mg/kg every 2 weeks, up to 12 cycles pre- and postoperatively
  Other Names: Avastin

SUMMARY:
This open-label, single arm, multicenter study evaluated the resection rate in participants with colorectal cancer and previously untreated unresectable liver-only metastases after adding bevacizumab to 5-FU based doublet chemotherapy in the neoadjuvant setting. Participants receive standard 5-FU based chemotherapy plus Avastin bevacizumab 5 milligrams per kilogram (mg/kg) every 2 weeks for a maximum of 12 cycles combined pre- and postoperatively, unless they experienced progressive disease or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Adult Chinese participants, 18-75 years of age
* Histologically confirmed adenocarcinoma in colon or rectum with primary lesion surgically removed
* Previously untreated unresectable liver-only metastases
* Liver lesions determined to be unresectable by multidisciplinary team (MDT, consisting of experienced hepatic surgeons, medical oncologist and radiologist).
* No previous treatment against liver metastases, including chemotherapy, surgery, radiotherapy, Transarterial chemoembolisation therapy (TACE) and target therapy
* Adequate hematological, renal and hepatic function
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Life expectancy greater than (>) 3 months

Exclusion Criteria:

* The relapse has occurred within 6 months of completion of the adjuvant treatment
* Expected impossible to achieve complete resection (R0 resection) and/or gain 30% residual liver volume even with responsive neoadjuvant therapy
* Participant cannot tolerate the surgery
* Other malignancies in the past 5 years, except for curatively treated basal cell carcinoma of the skin and/or in situ carcinoma of the cervix
* Any extrahepatic metastases and/or recurrence of the primary tumor
* Any residual toxicity from previous chemotherapy (except alopecia) of National Cancer Institute Common Toxicity Criteria (NCI CTC) v.4.0 grade 2
* Hypertension crisis or encephalopathy
* Pregnant or lactating women
* Clinically significant cardiovascular disease
* Evidence of bleeding diathesis or coagulopathy
* Current or recent (within 10 days of study drug initiation) use of full dose of aspirin, clopidrogel or warfarin
* History or evidence of Central Nervous System (CNS) disease (for example, primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of stroke)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-10-16 (Actual); Primary Completion 2015-04-04 (Actual); Study Completion 2016-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- China (7):
  - Beijing Cancer Hospital, Beijing
  - Sun Yet-sen University Cancer Center, Guangzhou
  - The Second Affiliated Hospital of Zhejiang University College, Hangzhou
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin
  - Zhongshan Hospital Fudan University, Shanghai
  - Liaoning cancer Hospital & Institute, Shenyang
  - Xiehe Hospital, Tongji Medical College Huazhong University of Science & Technology, Wuhan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Protocol did not specify any particular 5-Flurouracil (5-FU) based doublet chemotherapy regimen. The choice of 5-FU based doublet chemotherapy was as per standard of practice and the dosage of 5-FU based doublet chemotherapy was as per product labels.
Groups:
- Bevacizumab: Participants received standard 5-Flurouracil (5-FU) based chemotherapy plus bevacizumab 5 milligrams per kilograms (mg/kg) intravenous infusion every two week cycle for a maximum of 12 cycles unless they experienced progressive disease, unacceptable toxicities or participant refusal.
Period: Overall Study
Arm/Group | Bevacizumab
Started | 50
Completed | 12
Not Completed | 38
Not completed — Withdrawal by Subject | 18
Not completed — Progressive Disease | 8
Not completed — Investigator Decision | 5
Not completed — Lost to Follow-up | 4
Not completed — Protocol Violation | 2
Not completed — Unspecified Reason | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants enrolled in the study.
Groups:
- Bevacizumab: Participants received standard 5-FU based chemotherapy plus bevacizumab 5 mg/kg intravenous infusion every two week cycle for a maximum of 12 cycles unless they experienced progressive disease, unacceptable toxicities or participant refusal.
Arm/Group | Bevacizumab
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (9.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 39

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Complete Resection (R0 Resection)
Description: R0 resection was defined as complete resection confirmed by pathology after pre-operative chemotherapy plus bevacizumab. Participants with R0 resections based on assessments performed at time of surgery, 48 hours post-surgery and 4 and 12 weeks after surgery were reported.
Time Frame: At time of surgery (up to 28 weeks), 48 hours post-surgery and 4 and 12 weeks after surgery (up to 40 weeks)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 50
percentage of participants | 30.0 [17.9 to 44.6]

2. Secondary Outcome: Percentage of Participants Achieving Incomplete Tumor Resection (R1 Resection)
Description: R1 resection was defined as achievement of incomplete tumor resection with microscopic involvement of a margin after pre-operative chemotherapy plus bevacizumab, as confirmed by pathology. Participants with R1 resections based on assessments performed at time of surgery, 48 hours post-surgery and 4 and 12 weeks after surgery were reported.
Time Frame: At time of surgery (up to 28 weeks), 48 hours post-surgery and 4 and 12 weeks after surgery (up to 40 weeks)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 50
percentage of participants | 0.0 [0.0 to 7.1]

3. Secondary Outcome: Percentage of Participants Achieving Objective Response
Description: Objective response rate was defined as the percentage of participants who achieved either Partial Response (PR) or Complete Response (CR) per Response Evaluation Criteria In Solid Tumors (RECIST) version (v) 1.1. This is defined as the best response recorded from the start of trial treatment until disease progression (or death). CR was defined as complete disappearance of all target lesions and non-target disease, with the exception of nodal disease. All nodes, both target and non-target, must decrease to normal (short axis less than [<] 10 mm). No new lesions. PR was defined as greater than or equal to [≥] 30 percent (%) decrease under baseline of the sum of diameters of all target lesions. The short axis was used in the sum for target nodes, while the longest diameter was used in the sum for all other target lesions. No unequivocal progression of non-target disease. No new lesions.
Time Frame: Screening until disease progression or death until data cutoff on 12 May 2016 (up to approximately 3.5 years overall)
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 50
percentage of participants | 30.0 [17.9 to 44.6]

4. Secondary Outcome: Number of Participants With Disease Progression or Relapse or Death
Description: According to RECIST v1.1 Progressive Disease is defined as a 20 % or greater increase in the sum of the longest diameter of measured lesions (target lesions) taking as reference the smallest lesion diameter recorded since the treatment started or appearance of one or more new non-target lesions.
Time Frame: Screening until disease progression or death until data cutoff on 12 May 2016 (up to approximately 3.5 years overall)
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 50
participants | 28

5. Secondary Outcome: Progression Free Survival (PFS)
Description: Progressive Disease is defined as a 20% or greater increase in the sum of the longest diameter of measured lesions (target lesions) taking as reference the smallest lesion diameter recorded since the treatment started or appearance of one or more new non-target lesions. PFS was defined as the time from initiation of study treatment to disease progression, as determined by the investigator using RECIST v1.1 criterion, or relapse after resection of liver metastases or death from any cause. Kaplan-Meier curves were used to display PFS.
Time Frame: Screening until disease progression or death until data cutoff on 12 May 2016 (up to approximately 3.5 years overall)
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 50
months | 12.06 [6.70 to 13.31]

6. Secondary Outcome: Percent Probability (PP) of Being Alive and Progression Free at Months 3, 6, 9, 12, 15, and 18
Description: Progressive Disease is defined as a 20% or greater increase in the sum of the longest diameter of measured lesions (target lesions) taking as reference the smallest lesion diameter recorded since the treatment started or appearance of one or more new non-target lesions. PFS was defined as the time from initiation of study treatment to disease progression, as determined by the investigator using RECIST v1.1 criterion, or relapse after resection of liver metastases or death from any cause. The probability was estimated by Kaplan Meier curve analysis.
Time Frame: Months 3, 6, 9, 12, 15, and 18
Population: ITT population; Number of participants analyzed equals (=) number of participants who had surgery.
Measure: Number (95% Confidence Interval); unit: PP of being alive and progression free
Arm/Group | Bevacizumab
Number analyzed (Participants) | 17
PP of being alive and progression free
  3 Months | 97.7 [84.9 to 99.7]
  6 Months | 76.4 [59.4 to 87.0]
  9 Months | 59.5 [40.8 to 74.0]
  12 Months | 51.5 [32.6 to 67.5]
  15 Months | 30.0 [14.0 to 47.9]
  18 Months | 21.4 [8.1 to 38.9]

7. Secondary Outcome: Number of Participants With Disease Relapse or Death
Time Frame: Screening until disease progression or death until data cutoff on 12 May 2016 (up to approximately 3.5 years overall)
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 50
participants | 20

8. Secondary Outcome: Disease Free Survival (DFS)
Description: Disease Free Survival (DFS) was defined as the time from complete resection of liver metastases to disease relapse or death, for participants who achieve complete resection after pre-operative treatment with standard 5-FU based doublet regimen plus bevacizumab.
Time Frame: Complete resection date up to disease relapse or death until data cutoff on 12 May 2016 (up to approximately 3.5 years)
Population: ITT population; Here, number of participants analyzed = participants who underwent study specified surgery. Participants who underwent surgery but did not achieve complete resection were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 17
months | 8.48 [1.84 to 10.09]

9. Secondary Outcome: Percent Probability Of Being Alive and Disease Free at Months 3, 6, 9, and 12
Time Frame: Months 3, 6, 9, and 12
Population: ITT population
Measure: Median (95% Confidence Interval); unit: PP of being alive and disease free
Arm/Group | Bevacizumab
Number analyzed (Participants) | 50
PP of being alive and disease free
  3 Months | 80.0 [40.9 to 94.6]
  6 Months | 70.0 [32.9 to 89.2]
  9 Months | 40.0 [12.3 to 67.0]
  12 Months | 20.0 [3.1 to 47.5]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the date of Screening until data cutoff on 12 May 2016 (up to approximately 3.5 years overall)
Arm/Group | Bevacizumab
Serious Adverse Events (participants affected / at risk) | 4/50
Other Adverse Events (participants affected / at risk) | 26/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=50)
Abdominal infection (Infections and infestations) | 1
Scrotal infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=50)
Alanine aminotransferase increased (Investigations) | 7
Aspartate aminotransferase increased (Investigations) | 7
Neutrophil count decreased (Investigations) | 7
White blood cell count decreased (Investigations) | 5
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 4
Injection site reaction (General disorders) | 7
Hypertension (Vascular disorders) | 11
Bone marrow failure (Blood and lymphatic system disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.